CLINICAL TRIAL: NCT04057287
Title: Risk Factors of Liver Fibrosis Among First Degree Relatives of Patients With NASH Related Cirrhosis (NRC).
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-NRC-01
Record Dates: First submitted 2019-06-13; First posted 2019-08-15 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Liver Cirrhoses

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genetic markers like PNPLA3,TM6SF2,SAMM50, PARVB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NASH related Cirrhosis
  Interventions: Other: No intervention
- Healthy Controls
  Interventions: Other: No intervention
- First Degree Relatives of NASH related Cirrhosis
  Interventions: Other: No intervention
- HBV Disease Control
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The study aim to identify the risk factors of liver fibrosis among first degree relatives. This study consists of 2 parts (Cross Sectional and Case Control Study).

Part 1: The first primary objective will be achieved by following study design. Study population: First degree relatives of NRC. Study design: A Cross Sectional Study

Part 2 The second Primary objective will be achieved by following study design. Study design: A Case Control Study

Study population:

Case: NASH related Cirrhosis patients Control-1: Healthy Control. Control-2: HBV Disease Control Study period: 3 Years

All the patients diagnosed with NASH cirrhosis attending Institute of Liver and Biliary Sciences OPD/IPD will be enrolled. An informed consent will be taken. Complete details of the subject will be taken. The data will be collected on socio-demographic by (socio-demographic questionnaire), alcohol by AUDIT-C (Alcohol Use Disorders Identification Test), Tobacco by FTND (Fagerstrom Test Nicotine Dependence), physical activity by IPAQ (International Physical Activity Questionnaire), Diet by FFQ (Food Frequency Questionnaire), physical measurement & all the comorbidities.

Blood will be collected and analyzed for Platelets, PT/INR, Serum Creatinine, LFT, FBS, HOMA-IR, Lipid Profile, HBsAg, AntiHBs, Anti HBc, Anti HCV, Anti HAV, IgM anti HAV, IgM anti HEV, auto-Immune markers, Ceruloplasmin, Transferrin, S.Ferritin, Alpha1antitrpsin and genetic markers.

The stool will be collected and analyzed for gut microbiota profiling.

DETAILED DESCRIPTION:
The data will be collected on socio-demographic by (socio-demographic questionnaire), alcohol by AUDIT-C (Alcohol Use Disorders Identification Test), Tobacco by FTND (Fagerstrom Test Nicotine Dependence), physical activity by IPAQ (International Physical Activity Questionnaire), Diet by FFQ (Food Frequency Questionnaire), 24-hour dietary recall method, physical measurement & all the comorbidities.

Blood will be collected and analyzed for CBC, LFT, KFT, PT/INR, FBS, HOMA-IR, Lipid Profile, HBsAg, AntiHBs, Anti HBc, Anti HCV, Anti HAV, IgM anti HAV, IgM anti HEV, auto-Immune markers, Ceruloplasmin, Transferrin, S.Ferritin, Alpha1antitrpsin and genetic markers.

The stool will be collected and analyzed for gut microbiota profiling. Controlled Attenuation Parameter and liver stiffness will be measured by using transient elastography. Ultrasound abdomen will be done First degree relatives of indexed patients will be enrolled. First degree relatives who will not accompanying the indexed subject will be contacted telephonically and will be requested to participate in the study.

The data on first degree relative will be collected on similar parameter as of the indexed patient. This will be a cross sectional study.

For each case, 1 healthy controls will be taken. Healthy Control will be identified from the OPD/IPD of ILBS. Liver transplant donors, hospital volunteers, Blood Donors, healthy attendants who are accompanying other patients of different specialties will be enrolled. An informed consent will be taken. The data will be collected on similar parameter as of the indexed patient. This will be case control study.

We will also have disease control (HBV control) for each case enrolled. Subject suffering from Hepatitis B virus related liver cirrhosis will be included as disease control. For each case, 1 disease control will be included. Disease Control will be identified from the OPD/IPD of ILBS. An informed consent will be taken. The data will be collected on similar parameter as of the indexed patient.

Genetic markers and stool microbiota profiling will be done in 30% of the subsets of sample i.e NASH related Cirrhosis, First Degree Relatives, Healthy Control and HBV Disease control.

ELIGIBILITY:
Inclusion Criteria for NASH related Cirrhosis (Group 1-Index Case)

1. Age ≥18 yrs
2. Diagnosed cases of NASH with Cirrhosis.

Exclusion Criteria for NASH related Cirrhosis (Group 1)

1. Acute on Chronic Liver Failure
2. Patients with HBV, HCV, Wilson's, Hemochromatosis, alpha 1 antitrypsin deficiency, primary biliary cirrhosis).
3. Patient on treatment with amiodarone or methotrexate.
4. Patient with any malignancies
5. Patient on chemotherapy

Inclusion Criteria for First Degree Relatives (Group 2)

1. Age ≥8 yrs
2. All the first degree relatives of index case.

Exclusion Criteria for First Degree Relatives (Group 2)

1. Alcohol intake

Inclusion Criteria for Healthy Control (Group 3)

1. Age ≥18 yrs
2. Subjects with no history of any known liver disease
3. Non-Alcoholic
4. Matched with Age (+/- 5 yrs.) and Gender

Exclusion Criteria for Healthy Control (Group 3)

1. None

Inclusion Criteria for HBV Disease Control (Group 4)

1. Age ≥18 yrs
2. HBV Cirrhosis
3. Matched with Age (+/- 5 yrs.) and Gender

Exclusion Criteria for HBV Disease Control (Group 4)

1. Patient with any malignancies
2. HBV related Liver Fibrosis (≤ F3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NASH related Cirrhosis ( Group 1-Index Cases), First Degree Relatives of index case (Group 2), Healthy Controls (Group 3) HBV Disease Controls (Group 4)
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity-related risk factors as assessed using the International Physical Activity Questionnaire (IPAQ) between NASH related cirrhosis and their First Degree Relatives. | Day 0
Physical activity-related risk factors as assessed using the International Physical Activity Questionnaire (IPAQ) between NASH related cirrhosis and Healthy Control group. | Day 0
Dietary risk factors as captured by Food Frequency Questionnaire (FFQ) & 24 hour dietary recall method between NASH related cirrhosis and their First Degree Relatives. | Day 0
Dietary risk factors as captured by Food Frequency Questionnaire (FFQ) & 24 hour dietary recall method between NASH related cirrhosis and Healthy Control group | Day 0
Difference in microbiota profiling as done by 16s RNA sequencing technique between NASH related cirrhosis and their First Degree Relatives. | Day 0
Difference in microbiota profiling as done by 16s RNA sequencing technique between NASH related cirrhosis and Healthy Control group | Day 0
Genetic Single Nucleotide Polymorphism (SNP's) and Metabolic parameters in NASH related Cirrhosis patients and their 1st degree relatives. | Day 0
Genetic Single Nucleotide Polymorphism (SNP's) and Metabolic parameters in NASH related Cirrhosis patients and Healthy Control group. | Day 0
Metabolic syndrome as risk factors between NASH cirrhosis and their First Degree Relatives. | Day 0
Metabolic syndrome as risk factors between NASH cirrhosis and healthy Control | Day 0

SECONDARY OUTCOMES:
Proportion of Liver fibrosis among first degree relatives of patients with NASH related Cirrhosis. | Day 0
Physical activity-related risk factors as assessed using the International Physical Activity Questionnaire (IPAQ) between NASH related cirrhosis and HBV disease control. | Day 0
Dietary risk factors as captured by Food Frequency Questionnaire (FFQ) and 24 hours dietary recall method between NASH related cirrhosis and HBV disease control. | Day 0
Difference in microbiota profiling as done by 16s RNA sequencing technique between NASH related cirrhosis and HBV disease control. | Day 0
Genetic Single Nucleotide Polymorphism (SNP's) and Metabolic parameters in NASH related Cirrhosis patients and HBV disease control. | Day 0
Metabolic syndrome as risk factors between NASH cirrhosis and HBV Cirrhosis | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ankit Bhardwaj, Masters-CR, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided